CLINICAL TRIAL: NCT01945112
Title: Prevention Trial Assessing Paper-Tape in Endurance Distances II (Pre-TAPED II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Resurrection Medical Center (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 28548
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Blister of Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paper Tape (Experimental): Paper tape will be applied to study participants' blister prone areas or a randomly selected spot (if no blister history on that foot) - with untaped areas of the same foot as control.
  Interventions: Device: Paper Tape

INTERVENTIONS:
Device: Paper Tape — Applied to blister prone areas of the foot

SUMMARY:
Friction foot blisters are one of the most common and often debilitating complaints of all athletes, and hikers and runners in particular. Blistering rates in the literature of outdoor hikers range from 7%-54%. This study's aim is to build on Pre-TAPED I, and determine whether applying paper tape to the areas of the foot where blisters historically occur in endurance runners can prevent the incidence of friction blisters.

DETAILED DESCRIPTION:
Participants will be ultra-endurance athletes competing in Racing the Planet's 250 mile/7 day 4 Desert events in 2014 (Jordan, Gobi, Madagascar, and Atacama. A convenience sample will be used, with full consent signed before inclusion into the study, with participants being informed that study inclusion is entirely optional and will not affect medical care. Randomization will be conducted for each participant, a coin will be flipped to determine which foot is to be taped, heads - right foot, and tails, left foot. The non-taped foot will be used as a control. The runner's normal sock/shoe system will be used to reflect natural wilderness conditions. Participants will have demographic data collected prior to the race, including age, gender, country of origin, number of marathons run prior, pack weight, and sock type. The study endpoint occurs when a hot spot or blister develops on either the treated or untreated foot. Runners will be instructed to treat suspected blisters or hot spots as they normally would, and to inform the study administrators the same day for visual inspection and final questionnaire to determine if they develop blisters or hot spots, whether they applied or re-applied tape themselves, removed tape, and the reasons for these actions.

Participants will have tape applied to area(s) prone to blister on 1 foot, if no blister history, 1 area will be randomly assigned. The tape will be left on the selected foot until a blister or hot spot develops on either foot or the end of the race, whichever comes first. At that point, the study is over and the participant can continue or stop taping at their choice. If participants are prone to blisters or hot spots in particular areas, 1" paper tape applied to that site on trial foot. However, if the participant has no previous blister or hot spot experience, a site will be randomly assigned by picking a piece of paper out of a bag with the site written on a piece of paper (heel, toe, instep, head of 5th metatarsal). Therefore, a single participant can have more than 1 site on an individual foot.

ELIGIBILITY:
Inclusion Criteria:

Any runner who are enrolled in an RTP 4 deserts event, All runners who are 18-75 years old All runners who speak or read English. The study will be enrolling only those who speak or read English, so they can fully understand and have knowledgeable consent to the study enrollment protocols.

Exclusion Criteria:

Any blisters, broken blisters, or hot spots present on either foot at the time of initial taping as determined by visual foot inspection by a enrolling researcher.

The runner allergic to paper-tape.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Result] Lipman GS, Sharp LJ, Christensen M, Phillips C, DiTullio A, Dalton A, Ng P, Shangkuan J, Shea K, Krabak BJ. Paper Tape Prevents Foot Blisters: A Randomized Prevention Trial Assessing Paper Tape in Endurance Distances II (Pre-TAPED II). Clin J Sport Med. 2016 Sep;26(5):362-8. doi: 10.1097/JSM.0000000000000319. PMID 27070112

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: number of sites where tape was applied
Groups:
- Paper Tape on Right and No Tape on Left Foot; Paper Tape on Left and No Tape on Right Foot: Paper tape was applied to study participants' blister prone areas or a randomly selected spot (if no blister history on that foot) - with untaped areas of the same foot as control.
Period: Overall Study
Arm/Group | Paper Tape on Right and No Tape on Left Foot | Paper Tape on Left and No Tape on Right Foot
Started | 77; 153 number of sites where tape was applied (total number of sites where tape was applied) | 51; 87 number of sites where tape was applied (total number of sites where tape was applied)
Completed | 77; 153 number of sites where tape was applied | 51; 87 number of sites where tape was applied
Not Completed | 0; 0 number of sites where tape was applied | 0; 0 number of sites where tape was applied

BASELINE CHARACTERISTICS:
Groups:
- Paper Tape: Paper was applied to study participants' blister prone areas or a randomly selected spot (if no blister history on that foot) - with untaped areas of the same foot as control.
Arm/Group | Paper Tape
Number analyzed (Participants) | 128
Age, Continuous [Mean (Full Range); unit: years] | 39.3 [22 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 97

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Any Foot Blister in Taped or Untaped Area of the Foot
Description: Blister data were collected without regard to whether the foot was right or left.
Time Frame: within 7 days of application of tape
Measure: Count of Participants; unit: Participants
Groups:
- Paper Tape: Paper tape was applied to study participants' blister prone areas or a randomly selected spot (if no blister history on that foot) - with untaped areas of the same foot as control.
Arm/Group | Paper Tape
Number analyzed (Participants) | 128
Participants
  Blister anywhere | 106
  Blister in taped area | 30
  Blister in untaped area | 81

ADVERSE EVENTS:
Groups:
- Paper Tape on RIght Foot and No Tape on Left Foot; Tape on Left Foot and No Tape on Right Foot: Paper tape was applied to study participants' blister prone areas or a randomly selected spot (if no blister history on that foot) - with untaped areas of the same foot as control.
Arm/Group | Paper Tape on RIght Foot and No Tape on Left Foot | Tape on Left Foot and No Tape on Right Foot
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/51
Other Adverse Events (participants affected / at risk) | 0/77 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No